CLINICAL TRIAL: NCT05091060
Title: Erchonia and InnerScope, Pilot Evaluation of the Effect of the Erchonia® HLS™ for the Relief of Tinnitus Symptoms
Brief Title: Effect of the Erchonia® HLS™ for the Relief of Tinnitus Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-Tinnitus-Pilot
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Erchonia HLS (Experimental): 635 nanometers (nm) laser application
  Interventions: Device: Erchonia HLS

INTERVENTIONS:
Device: Erchonia HLS — 56 procedure administrations with the Erchonia® HLS™ administered by the subject at home: daily procedure administrations for 8 weeks.

SUMMARY:
This study is to see if applying red low-level laser light can help to reduce tinnitus symptoms

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the effectiveness of the Erchonia® HLS™, manufactured by Erchonia Corporation (the Company), in providing temporary relief of tinnitus symptoms in adults 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Subjective tinnitus
* Tonal tinnitus.
* Constant tinnitus on-going at least half the time over at least the past 6 months.
* Willing to abstain from other tinnitus-related treatments except prior hearing aid use throughout the study duration.
* Willing and able to refrain from activities or work involving excessive noise exposure without the use of effective hearing protection throughout study participation.
* 18 years of age or older
* Primary language is English

Exclusion Criteria:

* Objective tinnitus
* Atonal, pulsatile, intermittent, or occasional tinnitus
* Severe or profound hearing loss in one or both ears
* Current or prior surgically removed acoustic neuroma
* Consistent use of any of the following drugs known to cause or increase tinnitus (primarily ototoxins) within the past 30 days:

NSAIDS (motrin, naproxen, relafen, etc) aspirin (exceeding 300mg per day) and other salicylates Lasix and other "loop" diuretics "mycin" antibiotics such as vancomycin quinine and related drugs Chemotherapy agents such as cis-platin

* Acute or chronic vertigo/dizziness
* Ménière's disease
* Prior stapendectomy
* Prior mastoidectomy
* Auditory nerve tumor (acoustic neuroma), current or surgically removed in the past
* Active infection/wound/external trauma to the areas to be treated with the laser
* Medical, physical or other contraindications for, or sensitivity to, light therapy
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kathy Amos, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia HLS
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia HLS
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.25 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Score on the Tinnitus Handicap Inventory (THI).
Description: The Tinnitus Handicap Inventory (THI) is a 25-item questionnaire to assess how tinnitus affects an individual's life. Each question is responded to as 'yes' (4 points); 'sometimes' (2 points) or 'no' (0 points). The individual scores for the 25 questions are added to get a total THI score from 0 to 100. The higher the total THI score, the greater the negative impact tinnitus has on the individual's life. Change in total THI score is calculated as total THI score after the eight week procedure administration phase minus total THI score at baseline. A positive (+) change in total THI score indicates the negative impact of tinnitus on the individual's everyday life has worsened. A negative (-) change indicates the negative impact of tinnitus on the individual's everyday life has improved (lessened).
Time Frame: Baseline and 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erchonia HLS
Number analyzed (Participants) | 4
score on a scale | -24 (10.09)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Erchonia HLS
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT05091060/Prot_SAP_ICF_000.pdf